CLINICAL TRIAL: NCT00544726
Title: Rehabilitation for Patients With Pulmonary Arterial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rabin Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc074491ctl
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2007-10

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Rehabilitation
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Physical training
  Interventions: Behavioral: Physical training
- 2 (Placebo Comparator): No physical training
  Interventions: Behavioral: No training

INTERVENTIONS:
Behavioral: Physical training
  Arms: 1
Behavioral: No training
  Arms: 2

SUMMARY:
Patients suffering from pulmonary arterial hypertension (PAH) frequently remain symptomatic despite medical therapy. Symptoms include breathlessness, poor exercise capacity and reduced quality of life.

In many other serious heart or lung diseases it has been shown that physical rehabilitation improves patient's fitness and quality of life. In PAH there are no clear guidelines and in general physical activity has traditionally been discouraged, although evidence for this advice is lacking. Interesting research project in Germany showed significant benefit for in-patient rehabilitation in PAH patients.

In this study we will perform a controlled clinical study of out-patient rehabilitation of patients with PAH. We hypothesize that physical training of patients will result in increased exercise capacity and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

* All patients must satisfy current diagnostic criteria for pulmonary artery hypertension based on their historical right heart catheter data (within 4 years of study enrollment): Mean PAP >25mmHg at rest or >30mmHg with exercise, by a PCWP <= 15mmHg and by PVR >3 Wood Units.
* Willing and able to participate in 24 bi-weekly rehabilitation sessions, and medical follow-up.
* Stable dose of current PAH-specific medication for 3 months prior to enrollment.
* New York Heart Association (NYHA) Class II-III.
* Women of child-bearing age must demonstrate adequate contraception or undergo a pregnancy test.

Exclusion Criteria:

* Functional Class NYHA Class I or IV.
* PAH due to congenital heart disease, left heart disease, chronic lung diseases (VC or FEV1 < 60% of predicted) or chronic hypoxia.
* Acute intercurrent illness requiring hospital admission in the month proceeding screening.
* Any non-PAH medical condition likely to interfere with participation in rehabilitation, e.g. musculoskeletal disorders.
* Any uncontrolled or terminal non-PAH medical condition likely to interfere with completion of the study, according to the judgment of the study physician.
* Participation in another rehabilitation scheme within 6 months of enrollment in the study.
* Current participation in another clinical trial.
* Pregnancy or planned pregnancy during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Six minute walking distance | 3 months
New York Heart Association (NYHA) functional class | 3 months

SECONDARY OUTCOMES:
Echocardiographic parameters | 3 months
Quality of life as assessed by the SF-36 | 3 months
Performance in cardiopulmonary exercise test | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai R Kramer, MD, Study Director — Rabin Medical Center
Locations (1):
- Pulmonary Institute, Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Background] Mereles D, Ehlken N, Kreuscher S, Ghofrani S, Hoeper MM, Halank M, Meyer FJ, Karger G, Buss J, Juenger J, Holzapfel N, Opitz C, Winkler J, Herth FF, Wilkens H, Katus HA, Olschewski H, Grunig E. Exercise and respiratory training improve exercise capacity and quality of life in patients with severe chronic pulmonary hypertension. Circulation. 2006 Oct 3;114(14):1482-9. doi: 10.1161/CIRCULATIONAHA.106.618397. Epub 2006 Sep 18. PMID 16982941
- [Background] Nici L, Donner C, Wouters E, Zuwallack R, Ambrosino N, Bourbeau J, Carone M, Celli B, Engelen M, Fahy B, Garvey C, Goldstein R, Gosselink R, Lareau S, MacIntyre N, Maltais F, Morgan M, O'Donnell D, Prefault C, Reardon J, Rochester C, Schols A, Singh S, Troosters T; ATS/ERS Pulmonary Rehabilitation Writing Committee. American Thoracic Society/European Respiratory Society statement on pulmonary rehabilitation. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1390-413. doi: 10.1164/rccm.200508-1211ST. No abstract available. PMID 16760357
- [Derived] Fox BD, Kassirer M, Weiss I, Raviv Y, Peled N, Shitrit D, Kramer MR. Ambulatory rehabilitation improves exercise capacity in patients with pulmonary hypertension. J Card Fail. 2011 Mar;17(3):196-200. doi: 10.1016/j.cardfail.2010.10.004. Epub 2010 Dec 3. PMID 21362526